CLINICAL TRIAL: NCT01556139
Title: Evaluation of the Effectiveness of Respiratory Muscle Training by the Technique of Hypocapnia Hyperpnea (Spirotiger) in COPD and CHF Patients
Brief Title: Effectiveness of Respiratory Muscle Training by Spirotiger in Chronic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Mara Paneroni, Study Investigator, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Spirotiger
Record Dates: First submitted 2012-03-07; First posted 2012-03-16 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Congestive Heart Failure
Keywords: Endurance; exercise training; 6-min walking test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spirotiger (Experimental): Patients belonging to this group perform 20 sessions of usual training (cyclette and calisthenic exercises) and additional 20 sessions of a specific training for respiratory muscles with Spirotiger
  Interventions: Device: Spirotiger
- Control (No Intervention): Control group with a placebo device

INTERVENTIONS:
Device: Spirotiger — The Training group perform 20 sessions of a specific training with Spirotiger, a device allowing respiratory muscle training with isocapnic hyperpnea.
  The setting is the following:
  * volume/size of the breathing bag: 50% of the vital capacity (VC) and ventilation (VE= Tidal volume x respiratory rate) at 66% of the MVV aiming to reach 15 minutes of training without breaks. During the initial sessions, the patient can interrupt training every 5 minutes and recover.
  * increase in training: after 15 minutes of exercise VE is increased up to 75% of the MVV through modification of the volume of breathing bag or respiratory rate.
  At the end of 15 minutes of exercise, further increases in ventilation are 10% of each previous step.
  Arms: Spirotiger

SUMMARY:
The reduction in effort tolerance as result of a decreased efficiency in ventilation is common both in patients affected by COPD (McKenzie) and chronic heart failure (CHF) (Ribeiro, Frankenstein). One of the most common cause is the reduced respiratory muscle strength and endurance. Some studies have evaluated the effect of a specific training on the muscular strength both in pulmonary (Battaglia, Powell) and cardiac patients (Winkelmann, Chiappa). Moreover, only few studies investigated a specific training for such patients (Koppers, Sherer) because of the complicated equipment needed to prevent hypocapnia. Up to date, portable and economic systems for isocapnic hyperpnea have been developed for respiratory muscle training.

Primary aim of the study was to evaluate the effectiveness of the respiratory muscle training -by the technique of the isocapnic hyperpnea- on the effort tolerance and endurance in patients with COPD and CHF

Secondary aims were: A.to quantify the number of patients with deficit of respiratory muscles endurance and B.to verify different response of training between COPD and CHF patients

DETAILED DESCRIPTION:
All consecutive stable patients with diagnosis of COPD or CHF and normal MMSE, admitted in Foundation S. Maugeri in Lumezzane (Brescia, Italy) for routinary rehabilitation at Respiratory and Cardiac Rehabilitative Divisions are enrolled.

All patients who met the inclusion criteria (see above)are informed about the aim of the project, sign an informed consent and are enrolled in the study.

40 patients are enrolled. They are divided in two groups of 20 each (10 cardiac and 10 respiratory patients) named:

1. Spirotiger Group: these patients perform 20 sessions of usual training (cyclette and calisthenic exercises) and specific training (further 20 sessions) for respiratory muscles with SPIROTIGER
2. Control Group: these patients perform 20 sessions of usual training (cyclette and calisthenic exercises) and additional 20 sessions with a placebo device (Threshold)

ELIGIBILITY:
Inclusion Criteria:

* Ability to perform 6-min walking test.
* Emogas analysis at rest (with PaO2>60mmHg and PCO2<45 mmHg)
* Mini Mental State Examination (MMSE) > 25
* Absence of major events in the last month (i.e. respiratory exacerbation treated with antibiotic therapy, CHF unstabilization with administration of vasopressor drugs to support the cardiac pump).
* Maximum Voluntary Ventilation (MVV) as evaluation of endurance <90%.

Exclusion Criteria:

* Haemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in MVV | baseline and 20 days
  In patients with COPD and CHF,endurance is measured by Maximum Voluntary Ventilation Test (MVV)

SECONDARY OUTCOMES:
Changes in 6-min Walking test | baseline and 20 days
Changes in Spirometry parameters | baseline and 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Mara Paneroni, PT, Principal Investigator — Fondazione Salvatore Maugeri, Lumezzzane
Locations (1):
- Fondazione Salvatore Maugeri, Lumezzane, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Publication

REFERENCES:
- [Background] Ribeiro JP, Chiappa GR, Neder JA, Frankenstein L. Respiratory muscle function and exercise intolerance in heart failure. Curr Heart Fail Rep. 2009 Jun;6(2):95-101. doi: 10.1007/s11897-009-0015-7. PMID 19486593
- [Background] Frankenstein L, Nelles M, Meyer FJ, Sigg C, Schellberg D, Remppis BA, Katus HA, Zugck C. Validity, prognostic value and optimal cutoff of respiratory muscle strength in patients with chronic heart failure changes with beta-blocker treatment. Eur J Cardiovasc Prev Rehabil. 2009 Aug;16(4):424-9. doi: 10.1097/HJR.0b013e3283030a7e. PMID 19474739
- [Background] Battaglia E, Fulgenzi A, Ferrero ME. Rationale of the combined use of inspiratory and expiratory devices in improving maximal inspiratory pressure and maximal expiratory pressure of patients with chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2009 Jun;90(6):913-8. doi: 10.1016/j.apmr.2008.12.019. PMID 19480865
- [Background] Powell T, Williams EM. Inspiratory muscle training in adults with COPD. Respir Med. 2009 Aug;103(8):1239; author reply 1240-1. doi: 10.1016/j.rmed.2009.01.027. Epub 2009 Apr 11. No abstract available. PMID 19362808
- [Background] Winkelmann ER, Chiappa GR, Lima CO, Viecili PR, Stein R, Ribeiro JP. Addition of inspiratory muscle training to aerobic training improves cardiorespiratory responses to exercise in patients with heart failure and inspiratory muscle weakness. Am Heart J. 2009 Nov;158(5):768.e1-7. doi: 10.1016/j.ahj.2009.09.005. Epub 2009 Oct 2. PMID 19853695
- [Background] Chiappa GR, Roseguini BT, Vieira PJ, Alves CN, Tavares A, Winkelmann ER, Ferlin EL, Stein R, Ribeiro JP. Inspiratory muscle training improves blood flow to resting and exercising limbs in patients with chronic heart failure. J Am Coll Cardiol. 2008 Apr 29;51(17):1663-71. doi: 10.1016/j.jacc.2007.12.045. PMID 18436118
- [Background] Koppers RJ, Vos PJ, Boot CR, Folgering HT. Exercise performance improves in patients with COPD due to respiratory muscle endurance training. Chest. 2006 Apr;129(4):886-92. doi: 10.1378/chest.129.4.886. PMID 16608934
- [Background] Scherer TA, Spengler CM, Owassapian D, Imhof E, Boutellier U. Respiratory muscle endurance training in chronic obstructive pulmonary disease: impact on exercise capacity, dyspnea, and quality of life. Am J Respir Crit Care Med. 2000 Nov;162(5):1709-14. doi: 10.1164/ajrccm.162.5.9912026. PMID 11069801
- [Background] McKenzie DK, Butler JE, Gandevia SC. Respiratory muscle function and activation in chronic obstructive pulmonary disease. J Appl Physiol (1985). 2009 Aug;107(2):621-9. doi: 10.1152/japplphysiol.00163.2009. Epub 2009 Apr 23. PMID 19390004
- [Result] Paneroni M, Simonelli C, Saleri M, Trainini D, Fokom G, Speltoni I, Piaggi G, Ambrosino N, Vitacca M. Short-Term Effects of Normocapnic Hyperpnea and Exercise Training in Patients With Chronic Obstructive Pulmonary Disease: A Pilot Study. Am J Phys Med Rehabil. 2018 Dec;97(12):866-872. doi: 10.1097/PHM.0000000000000988. PMID 29927750